CLINICAL TRIAL: NCT04388774
Title: A Phase 2A Open-Label Study Evaluating the Safety and Efficacy of Low-Dose Ketamine in Children With ADNP Syndrome
Brief Title: Low-Dose Ketamine in Children With ADNP Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexander Kolevzon (Other)
Responsible Party: Sponsor-Investigator, Alexander Kolevzon, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-1253
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: ADNP Syndrome
Keywords: Ketamine; ADNP; Activity-Dependent Neuroprotector Protein; Chromosome Disorders; Chromosome Aberrations
MeSH Terms: conditions — Chromosome Disorders; Chromosome Aberrations | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): Total dose administration or 0.5 mg/kg of ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — A single 40-minute intravenous infusion

SUMMARY:
This is a Phase 2A, single dose, open-label study to evaluate the safety, tolerability, and efficacy of a low-dose, 40-minute infusion into the veins (intravenous infusion or "IV") of ketamine in children with ADNP syndrome (Activity-Dependent Neuroprotective Protein). The study team will enroll 10 participants, ages 5 to 12, at Mount Sinai. The study participation is expected to last 4 weeks and will include 5 scheduled clinic visits in order to complete safety monitoring, clinical assessments, and biomarker collection. At the conclusion of this study, the study team expects to demonstrate the safety and tolerability of low-dose ketamine in children with ADNP syndrome. Additionally, the study team anticipates identifying meaningful signals of efficacy in clinical outcome measures using RNA and DNA sequencing to analyze ADNP protein expression and DNA methylation profiles, a natural process by which methyl groups are added to the DNA to change its activity, in order to assess sensitivity to change with low-dose ketamine treatment and inform future phase 3 studies. Ketamine is not currently approved by the Food and Drug Administration to treat this syndrome, but it is approved for use in children in other situations, for example in anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 12 years old (inclusive) at the time of informed consent;
* Has a diagnosis of ADNP syndrome, confirmed by genetic testing prior to subject randomization;
* Has a Clinical Global Impression-Severity score of 4 (moderately ill) or greater at screening;
* Any concomitant medication, including anti-epileptic and/or behavioral medications, supplements, and special diets, must be at a stable dose for at least 4 weeks before;
* Has an English-speaking caregiver capable of providing informed consent and able to attend all scheduled study visits, oversee the administration of study drug, and provide feedback regarding the subject's behavior and other symptoms as described in the protocol;
* Provide assent to the protocol (when applicable);
* Has a caregiver who will agree not to post any of the subject's personal medical data related to the study or information related to the study on any website or social media site (e.g., Facebook and Twitter) until they have been notified that the study is completed.
* Age-specific blood pressure parameters for inclusion in the study will be based on established guidelines.

Exclusion Criteria:

* Has a concomitant disease (e.g., gastrointestinal, renal, hepatic, endocrine, respiratory, or cardiovascular system disease) or condition or any clinically significant finding at screening that could interfere with the conduct of the study or that would pose an unacceptable risk to the subject in this study;
* Has clinically significant lab abnormalities or vital signs at the time of screening (e.g., alanine aminotransferase or aspartate aminotransferase >2.5 × upper limit of normal; total bilirubin or creatinine >1.5 × upper limit of normal). Re-testing of safety labs is allowed;
* Hypertension that is not well controlled (systolic BP >130-140 mm Hg or diastolic BP >85-95 mm Hg depending on age);
* A blood pressure reading over 160/90 or two separate readings over 140/90 at screening or baseline visits;
* Thyroid impairment, as reflected by a TSH > 4.2 mU/L;
* Cardiac disease, as reflected by an EKG that is abnormal and of concern for cardiac disease;
* Has had changes in his/her medication regimen within the previous month;
* Has a history of uncontrollable seizure disorder or seizure episodes within 1 month of screening;
* Has a history of suicidal behavior or considered by the investigator to be at high risk of suicide;
* Has a current or past history of psychotic symptoms;
* Has enrolled in any clinical trial or used of any investigational agent, device, and/or investigational procedure within the 30 days before screening or does so concurrently with this study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten participants were screened, and all met criteria for inclusion and were enrolled between August 2020 and May 2021.
Groups:
- Ketamine: Single-dose (0.5 mg/kg) infused intravenously over 40 minutes
Period: Overall Study
Arm/Group | Ketamine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.50 (2.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 2
  White | 8
Developmental quotient [Mean (Standard Deviation); unit: quotient] — A development quotient (DQ) is a numerical indicator of a child's growth to maturity across a range of psychosocial competencies.
  Developmental quotient (DQ) is calculated as follows: DQ = [developmental age (DA)] divided by chronological age (CA) ×100
  quotient
    VDQ - verbal developmental quotient | 26.71 (15.33)
    NVDQ - nonverbal developmental quotient | 31.28 (16.13)
    FSDQ - full scale developmental quotient | 28.81 (15.42)
Number of Participants with ASD [Count of Participants; unit: Participants] — ASD: autism spectrum disorder
  Participants | 4
Number of Participants with ADHD [Count of Participants; unit: Participants] — ADHD: attention deficit/hyperactivity disorder
  Participants | 7
Genetic mutation [Count of Participants; unit: Participants]
  Frameshift | 6
  Nonsense | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Description: Number of Participants with an adverse event as defined by the Systematic Longitudinal Assessment of Adverse Events (SLAES) which is a comprehensive form that assesses medical and behavioral conditions that were present at screening and/or baseline. Conditions are considered treatment emergent if their severity increased significantly after the participant had taken at least one dose of the study treatment. Treatment emergent adverse events will be tracked considered in the adverse event safety analysis. Severity of adverse events are categorized as mild, moderate, severe, life-threatening, or resulting in death and the treating physician indicates if the adverse event was related or unrelated to study drug.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine
Number analyzed (Participants) | 10
Participants | 9

2. Secondary Outcome: Aberrant Behavior Checklist
Description: Changes in scale at week 1 compared to baseline. Aberrant Behavior Checklist is a behavior rating scale for the assessment of treatment effects. Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). Subscales from 0-45 for Irritability; 0-48 for Social Withdrawal and Hyperactivity; from 0-21 for Stereotypy; and 0-12 for In Speech , with total scale from 0 to 48, with higher score indicating worse health outcomes.
Time Frame: Baseline, Week 1
Population: Each participant had one caregiver provide rated assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregiver Rated Assessment at Baseline: Caregiver rated assessments at baseline
- Caregiver Rated Assessment at 1 Week: Caregiver rated assessments at 1 week
Arm/Group | Caregiver Rated Assessment at Baseline | Caregiver Rated Assessment at 1 Week
Number analyzed (Participants) | 10 | 10
score on a scale
  Irritability | 20.5 (13.33) | 10.9 (10.6)
  Social withdrawal | 9.9 (8.96) | 4.2 (4.96)
  Motor stereotypies | 7.8 (5.31) | 4.5 (3.66)
  Hyperactivity | 24.5 (14.66) | 16.2 (13.35)
  Inappropriate speech | 3.6 (2.88) | 3.3 (2.21)

3. Secondary Outcome: Anxiety, Depression and Mood Scales (ADAMS)
Description: The ADAMS is a parent/caregiver-completed measure and consists of 28 items, grouped into five subscales (Manic/Hyperactive Behavior, Depressed Mood, Social Avoidance, General Anxiety, Obsessive Behavior), and scored on a four-point Likert scale that combines frequency and severity ratings from 0-3. Subscales range - Hyperactivity 0-15; Depressed 0-21; Social Avoidance 0-21; General anxiety 0-21; OCD 0-9. Scores are not summed. Higher score indicates poorer health outcomes.
Time Frame: Baseline and Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregiver Rated Assessment Week 1: caregiver rated assessments at week 1
Arm/Group | Caregiver Rated Assessment at Baseline | Caregiver Rated Assessment Week 1
Number analyzed (Participants) | 10 | 10
score on a scale
  Hyperactivity | 10.1 (4.23) | 6.7 (3.5)
  Depressed | 2.6 (3.31) | 2.1 (2.69)
  Social avoidance | 6.1 (4.23) | 3.5 (3.47)
  General anxiety | 6.3 (5.96) | 4.3 (4.74)
  Obsessive/compulsive | 2.5 (2.01) | 1.6 (1.51)

4. Secondary Outcome: Repetitive Behavior Scale-Revised (RBS-R)
Description: Change in repetitive behaviors at weeks 1 compared to baseline. RBS-R subscales - Stereo 0-18; Self injury 0-24; Compulsive 0-24; Ritualistic 0-18; Sameness 0-33; Restricted 0-12. Total scale range from 0 to 126 with higher score indicating worse health outcomes.
Time Frame: Baseline, Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Rated Assessment at Baseline | Caregiver Rated Assessment at 1 Week
Number analyzed (Participants) | 10 | 10
score on a scale
  Stereotyped | 6.6 (3.31) | 5.1 (4.93)
  Self-injury | 5.9 (4.79) | 4.2 (3.49)
  Compulsive | 3.7 (2.75) | 2.2 (1.87)
  Ritualistic | 2.9 (3.63) | 2.9 (2.38)
  Sameness | 5.6 (6.33) | 4.3 (5.46)
  Restricted | 3.9 (3.14) | 3.6 (2.37)
  Overall | 28.6 (17.56) | 22.3 (14.28)

5. Secondary Outcome: Clinical Global Impressions - Improvement Scale (CGI-I)
Description: Changes in scale at weeks 2, and 4 compared to baseline. Clinical Global impressions - Improvement Scale is anchored to symptoms of ADNP syndrome for the assessment of treatment effects. CGI-I total score from 1 to 7 point scale, with higher score indicating worse health outcomes.
Time Frame: Baseline, Week 2, and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 10
score on a scale
  Baseline | 0 (0)
  Week 2 | 1.5 (0.53)
  Week 4 | 1.0 (0.52)

6. Secondary Outcome: Childrens Sleep Habits Questionnaire
Description: Change in sleep habits at week 1 compared to baseline. Full scale from 0 to 110, with higher score indicating worse health outcomes.
Time Frame: Baseline, Week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Rated Assessment at Baseline | Caregiver Rated Assessment at 1 Week
Number analyzed (Participants) | 10 | 10
units on a scale | 2.83 (0.75) | 2.93 (0.82)

7. Secondary Outcome: Peabody Picture Vocabulary Test and Expressive Vocabulary Test
Description: Expressive and receptive language assessed by Peabody Picture Vocabulary Test and Expressive Vocabulary Test at Day 1, Weeks 1, 2, and 4. Full scale from 40 to 160, with higher score indicating better health outcomes.
Time Frame: Baseline, Week 1, Week 2, and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 10
score on a scale
  Baseline, Day 1 | 50.9 (13.40)
  Week 1 | 52.8 (17.38)
  Week 2 | 51.5 (13.87)
  Week 4 | 50.9 (15.29)

8. Secondary Outcome: Proportion of Target-First Trials Saccades
Description: Change at Day 1 and Week 1 as compared to baseline using computerized eye tracking to record where the subject is looking during an activity in which the subject will see a video of a person with two objects, turning her head towards one of the objects, the target.
  Mean proportion of trials in which participants made saccades to the target before the distractor.
Time Frame: Baseline, Day 1, Week 1
Population: Not every trial was valid. Eye tracking data were successfully collected from nine participants for the Joint Attention task, but only four participants had >25% valid trials at all three time points and were included in analysis.
Measure: Mean (Standard Deviation); unit: proportion of target-first saccades
Units Other Than Participants: Trials
Arm/Group | Ketamine
Number analyzed (Participants) | 4
Number analyzed (Trials) | 48
proportion of target-first saccades
  Baseline: number analyzed (Trials) | 31
  Baseline | 0.53 (0.14)
  Day 1: number analyzed (Trials) | 21
  Day 1 | 0.75 (0.17)
  Week 1: number analyzed (Trials) | 25
  Week 1 | 0.70 (0.14)

9. Secondary Outcome: Latency to First Saccade
Description: Change at week 1, week 2, and week 4 as compared to baseline using computerized eye tracking to record where the subject is looking during an activity in which the subject will see different social and non-social stimuli.
  Latency to first saccade to the target
Time Frame: Baseline, Day 1, Week 1
Population: Eye tracking data were successfully collected from nine participants for the Joint Attention task, but only four participants had >25% valid trials at all three time points and were included in analysis.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Ketamine
Number analyzed (Participants) | 4
ms
  Baseline | 2319.38 (1202.34)
  Day 1 | 2089.96 (754.70)
  Week 1 | 1674.18 (301.93)

10. Secondary Outcome: Proportion of Target-Dwelling
Description: Change at Day 1 and Week 1 as compared to baseline using computerized eye tracking to record where the subject is looking during an activity in which the subject will see different social and non-social stimuli.
  Proportion of time participants spent dwelling on the target versus distractor.
Time Frame: Baseline, Day 1, Week 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: proportion of time
Arm/Group | Ketamine
Number analyzed (Participants) | 4
proportion of time
  Baseline | 0.51 (0.19)
  Day 1 | 0.59 (0.13)
  Week 1 | 0.66 (0.11)

11. Secondary Outcome: Electrophysiology Recording
Description: Electroencephalographic recordings to measure Auditory Event Related Potentials at baseline, week 1, week 2, and week 4.
  In separate blocks, participants heard a 500-ms click at either a stimulation rate of 40 or 20 Hz. Click trains were presented 150 times each, with an intertrial interval of 50 ms, at approximately 60 db.
  Higher number indicates higher amplitude neural response to auditory stimuli.
Time Frame: Baseline, Week 1, Week 2, and Week 4
Population: participants with fewer than five wavelets at any time point were excluded
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Ketamine
Number analyzed (Participants) | 10
ms
  20-Hz Baseline: number analyzed (Participants) | 8
  20-Hz Baseline | 0.18 (0.06)
  20-Hz Week 1: number analyzed (Participants) | 8
  20-Hz Week 1 | 0.15 (0.05)
  20-Hz Week 2: number analyzed (Participants) | 8
  20-Hz Week 2 | 0.18 (0.06)
  20-Hz Week 4: number analyzed (Participants) | 8
  20-Hz Week 4 | 0.19 (0.11)
  40-Hz Baseline: number analyzed (Participants) | 7
  40-Hz Baseline | 0.19 (0.03)
  40-Hz Week1: number analyzed (Participants) | 7
  40-Hz Week1 | 0.26 (0.09)
  40-Hz Week 2: number analyzed (Participants) | 7
  40-Hz Week 2 | 0.18 (0.06)
  40-Hz Week 4: number analyzed (Participants) | 7
  40-Hz Week 4 | 0.20 (0.06)

12. Secondary Outcome: Vineland Adaptive Behavior Scales
Description: Changes in scale at week 4 compared to baseline. Vineland Adaptive Behavior Scales measures adaptive functioning. Higher score indicating better health outcomes. Domain scores are standard scores - population mean 100 standard deviation 15.
  an overall composite score, it consists of three subscales: (a) communication (receptive, expressive, written), (b) socialization (interpersonal relationships, play and leisure, coping skills), and (c) daily living (person, domestic, community).
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregiver Rated Assessment at Week 4: Caregiver rated assessments at week 4
Arm/Group | Caregiver Rated Assessment at Baseline | Caregiver Rated Assessment at Week 4
Number analyzed (Participants) | 10 | 10
score on a scale
  Abc | 42.7 (13.9) | 44.0 (15.19)
  Comm | 32.6 (14.73) | 33.4 (15.53)
  Daily Living | 48.5 (14.45) | 49.2 (16.14)
  Social | 44.5 (15.62) | 46.8 (16.90)
  Motor | 51.5 (8.73) | 49.83 (4.58)

13. Secondary Outcome: Caregiver Strain Questionnaire (CGSQ)
Description: Caregiver Strain Questionnaire (CGSQ) is a 13 question tool, with a 5-point Likert scale ranging from Not at all (0) to Very much (4). Domains (Objective strain, Subjective externalized strain, Subjective internalized strain) are averaged scores, range from 0-4. Total score (Global score) is a sum of the three subdomains. Full scale range 0-12, higher score indicates more severe strain.
Time Frame: Baseline and Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Rated Assessment at Baseline | Caregiver Rated Assessment at 1 Week
Number analyzed (Participants) | 10 | 10
score on a scale
  Objective strain | 2.79 (1.11) | 2.45 (0.99)
  Subjective externalized strain | 2.18 (1.11) | 1.62 (0.69)
  Subjective internalized strain | 3.3 (1.15) | 2.7 (0.97)
  Global score | 8.27 (3.08) | 6.77 (2.32)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=10)
Elated/silly (Psychiatric disorders) | 5
Aggression (Psychiatric disorders) | 4
Fatigue (Nervous system disorders) | 4
Decreased appetite (General disorders) | 3
Anxiety (Psychiatric disorders) | 3
Increased appetite (General disorders) | 2
Restless (Psychiatric disorders) | 2
Increased fluid intake (General disorders) | 2
Nausea/vomiting (Gastrointestinal disorders) | 2
Moody/irritable (Psychiatric disorders) | 2
Dry mouth (General disorders) | 2
Gagging/reflux (Gastrointestinal disorders) | 1
Self-injury (Psychiatric disorders) | 1
Loose stool (Gastrointestinal disorders) | 1
Difficulty falling asleep (Nervous system disorders) | 1
Early morning wakening (Nervous system disorders) | 1
Limping with possible pain (Musculoskeletal and connective tissue disorders) | 1
Decreased fluid intake (General disorders) | 1
Distractibility (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Increased frustration (Psychiatric disorders) | 1
Oppositional (Psychiatric disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Agitation (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT04388774/Prot_000.pdf